CLINICAL TRIAL: NCT01085604
Title: Recurrent Low Back Pain:Linking Mechanisms to Outcomes
Status: Completed | Type: Observational
Sponsor: Drexel University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sheri Silfies, Associate Professor, Drexel University
Other Study IDs: K01HD053632T; K01HD053632 (NIH)
Record Dates: First submitted 2010-03-10; First posted 2010-03-12 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Low Back Pain
Keywords: low back pain; clinical instability; neuromuscular control; core stabilization; physical therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Low back pain: Individuals with current low back pain attributed to poor trunk neuromuscular control (clinical instability).
  Interventions: Other: Core Stabilization

INTERVENTIONS:
Other: Core Stabilization — The 8-week core stabilization program emphasizes use of specific local stabilizing muscles (transverse abdominis[TrA], lumbar multifidus[LM]) to restore active control and stability to the trunk. This program emphasizes training using isometric co-contractions and a progression (3 stages) based upon a motor learning paradigm.
  Stage 1: emphasizes neutral position of the spine and activation of the TrA and LM. Performance feedback is emphasized and monitored through observation and palpation.
  Stage 2: promotes maintenance the co-contraction while performing movements of the trunk and superimposing movements of the upper and lower extremities. Trunk conditioning is also emphasized (i.e., curl ups, quadruped leg/arm lifts and side support). Feedback is gradually reduced.
  Stage 3: emphasis on maintenance of the co-contraction while performing exercises on an unstable surface or during perturbation of the activity. Random practice patterns are used to enhance motor learning.

SUMMARY:
The purpose of this study is to determine if trunk neuromuscular control strategies are changed by therapeutic exercises emphasizing core stabilization.

Hypothesis: subjects with low back pain who demonstrate clinically meaningful improvements in function and pain will have significantly improved trunk motor control strategies.

Hypothesis: measures of trunk control will demonstrate 'construct-validity'. This will be tested using a known group method demonstrating:

* no significant change in motor control measures within the untreated, healthy control group.
* significant changes within the low back subjects who demonstrate clinically meaningful improvements.

DETAILED DESCRIPTION:
A growing body of evidence suggests that poor neuromuscular control of the lumbopelvic region is an important finding in a large number of patients with recurrent and chronic low back pain and may play a role in recurrence of symptoms. Despite findings of altered trunk motor control in individuals with low back pain, the neuromuscular strategies underlying these alterations have not been satisfactorily characterized. The aims of this study are to(1) identify which neural control strategies are altered following a rehabilitation program that emphasizes trunk control and stability using a motor learning approach and (2) provide preliminary evidence of a link between hypothesized mechanism and effectiveness for programs designed to improve trunk control.

ELIGIBILITY:
Inclusion criteria for healthy controls:

No history of low back is defined as:

1. no pain limiting performance of daily activities for greater than 3 days,
2. no pain for which they sought medical or allied health intervention.

Inclusion Criteria for individuals with a history of low back pain:

1. duration of the current episode of low back pain less than 3 months,
2. average pain intensity over past 2 weeks at least 3 on an 11 point (0 = no pain, 10 = worst pain ever) numeric pain rating scale,
3. no medical intervention for low back pain in last 6 months,
4. Oswestry disability score greater than 20%
5. a physical therapy diagnosis of clinical lumbar instability based upon specific examination findings.

Exclusion Criteria for both groups:

1. permanent structural spinal deformity (e.g., scoliosis)
2. history of spinal fracture or diagnosis of osteoporosis
3. diagnosis of inflammatory joint disease
4. signs of systemic illness or suspected non-mechanical LBP (i.e. spinal tumor or infection)
5. previous spinal surgery
6. frank neurological loss, i.e., weakness and sensory loss
7. history of neurologic disease that required hospitalization,
8. active treatment of another medical illness that would preclude participation in any aspect of the study or any lower extremity injury that would potentially alter trunk movement in standing
9. leg length discrepancy of greater than 2.5 cm.
10. pregnancy
11. vestibular dysfunction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic physical therapy clinic community
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2009-08; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Trunk Neuromuscular Control | Baseline, 8 weeks
  Using surface EMG, trunk kinematics and force plate parameters. Trunk motor control is characterized and compared between groups and pre/post intervention in the low back pain group.

SECONDARY OUTCOMES:
Oswestry Disability Index | Baseline, 8 weeks
  measure of functional limitations

CONTACTS AND LOCATIONS:
Overall Officials: Sheri P. Silfies, PT, PhD, Principal Investigator — Drexel University
Locations (2):
- United States (2):
  - Drexel University, Philadelphia, Pennsylvania
  - Optimum Physical Therapy Associates, West Chester, Pennsylvania

REFERENCES:
- [Result] Sung W, Abraham M, Plastaras C, Silfies SP. Trunk motor control deficits in acute and subacute low back pain are not associated with pain or fear of movement. Spine J. 2015 Aug 1;15(8):1772-82. doi: 10.1016/j.spinee.2015.04.010. Epub 2015 Apr 8. PMID 25862508
- [Result] Mehta R, Cannella M, Henry SM, Smith S, Giszter S, Silfies SP. Trunk Postural Muscle Timing Is Not Compromised In Low Back Pain Patients Clinically Diagnosed With Movement Coordination Impairments. Motor Control. 2017 Apr;21(2):133-157. doi: 10.1123/mc.2015-0049. Epub 2016 Aug 19. PMID 26623551